CLINICAL TRIAL: NCT05207488
Title: Gastrointestinal And Metabolic Effects From a Prebiotic, Lifting, and Aerobic iNtervention (GAMEPLAN)
Brief Title: Gastrointestinal And Metabolic Effects From a Prebiotic, Lifting, and Aerobic iNtervention
Acronym: GAMEPLAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21730
Record Dates: First submitted 2021-09-21; First posted 2022-01-26 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
Keywords: Gastrointestinal microbiota; Fructooligosaccharides; Exercise; Fiber; Prebiotic; Short-chain fatty acids; Glucose homeostasis; Body composition; Cognition
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — fructooligosaccharide; Exercise; maltodextrin

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled trial with a 6-week intervention period with two groups: 1) Exercise + Prebiotic and 2) Exercise + Placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is a double-blind, placebo-controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + Prebiotic (Experimental): The Exercise + Prebiotic intervention group will consume 10 g/d of fructo-oligosaccharides (FOS). Additionally, they will perform 6 wk. of supervised progressive multi-component exercise training consisting of moderate to vigorous aerobic and strength-based exercises (3x/wk).
  Interventions: Dietary Supplement: Fructooligosaccharides (FOS); Behavioral: Exercise
- Exercise + Placebo (Placebo Comparator): The Exercise + Placebo group will consume 10 g/d of a placebo (maltodextrin) powder every day. Additionally, they will perform 6 wk. of supervised progressive multi-component exercise training consisting of moderate to vigorous aerobic and strength-based exercises (3x/wk).
  Interventions: Behavioral: Exercise; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fructooligosaccharides (FOS) — FOS (NUTRAFLORA® P-95, Ingredion) supplements (10g/day) will be consumed daily mixed with water.
  Arms: Exercise + Prebiotic
Behavioral: Exercise — During the intervention period, all participants will perform 6 weeks of supervised progressive multi-component exercise training consisting of moderate to vigorous aerobic and strength-based exercises (3x/wk.).
Dietary Supplement: Placebo — Maltodextrin (Globe 18DE Maltodextrin, Ingredion) supplements (10g/day) will be consumed daily mixed with water.
  Other Names: Maltodextrin
  Arms: Exercise + Placebo

SUMMARY:
This study aims to determine the independent and combined effects of prebiotic fiber supplementation and exercise on the gut microbiome and human health.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-45 kg/m2
* Without physician diagnosed gastrointestinal or metabolic diseases
* Sedentary (< 30 minutes of moderate or high intensity exercise per week OR < 20 aggregate Godin-Shepard Leisure Time Physical Activity Questionnaire (GSLTQ; GodinLeisure) score)
* Fully vaccinated against COVID-19

Exclusion Criteria:

* Fasting blood glucose >126 mg/dL
* Blood pressure >160/100 mm Hg
* Physician diagnosed metabolic or gastrointestinal diseases or constipation
* Heart conditions that may pose risk during exercise
* Taking oral hypoglycemic agents or insulin
* Pregnant, breastfeeding or postmenopausal
* Smoke or consume > 2 alcoholic beverages/day, abuse drugs
* Have had > 5% weight change in the past month or > 10% change in the past year
* Have had any form of bariatric surgery or gallbladder removal
* Have taken antibiotics during the previous 3 months
* Unable to consume the experimental fiber

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Changes in gastrointestinal microbiota composition | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on the gastrointestinal microbiota compared to control by sequencing the V4 region of the 16S rRNA gene in fecal samples.
Changes in gastrointestinal microbial-derived metabolite concentrations | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on the concentration of short-chain fatty acids compared to control.

SECONDARY OUTCOMES:
Changes in fasting glucose | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on fasting glucose compared to control.
Changes in fasting insulin | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on fasting insulin compared to control.
Changes in body composition | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on body composition compared to control. This includes percentage of fat mass and lean mass.
Changes in body fat distribution | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on body fat distribution compared to control. This includes the weight of visceral fat and liver fat in kilograms.
Changes in cognition | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on relational memory, hippocampal function, interference control, and selective attention compared to control. Outcomes will be assessed with computer tasks and participants will be equipped with an electrode cap.

OTHER OUTCOMES:
Changes in lipid profiles | Baseline & 6-week mark
  Determine the impact of daily consumption of prebiotic combined with regular exercise on fasting lipid profiles including cholesterol and triglycerides compared to control.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No